CLINICAL TRIAL: NCT04562727
Title: Microwave Ablation Combined With Chemotherapy for Colorectal Liver Metastases： a Multicenter Cohort Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ping Liang (Other)
Responsible Party: Sponsor-Investigator, Ping Liang, Interventional ultrasound department, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S2020-266-01
Record Dates: First submitted 2020-09-06; First posted 2020-09-24 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Colorectal Carcinoma; Chemotherapy; Liver Metastases
Keywords: Microwave Ablation; Colorectal liver metastasis
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Only MWA (Experimental): Only preform MWA, chemotherapy isn't necessary
  Interventions: Drug: Chemotherapy
- MWA combined with perioperative chemotherapy (Active Comparator): MWA combined with perioperative chemotherapy. Chemotherapy was preformed before MWA and after MWA
  Interventions: Drug: Chemotherapy
- MWA combined with postoperative chemotherapy (Experimental): MWA combined with perioperative chemotherapy. Chemotherapy was preformed after MWA
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Chemotherapy — perioperative chemotherapy or postoperative chemotherapy
  Other Names: preoperative chemotherapy; postoperative chemotherapy

SUMMARY:
Colorectal cancer is the second deadliest malignant tumor worldwide, and liver is the most common site of hematogenic metastasis of Colorectal cancer. Surgery is an effective treatment for colorectal cancer with liver metastasis, however, only 10%-20% of patients with liver metastasis are feasible for radical surgical resection. Many single-center retrospective studies have demonstrated that thermal ablation for liver metastases is comparable to surgery. Chemotherapy can kill the microscopic cancer foci of the liver. The timing of ablation-related chemotherapeutic administration still needs to be explained.

The purpose of this study was to compare the clinical efficacy of thermal ablation or combined with perioperative chemotherapy and postoperative chemotherapy in the treatment of colorectal cancer with liver metastasis.

DETAILED DESCRIPTION:
Colorectal cancer is the second deadliest malignant tumor worldwide, and liver is the most common site of hematogenic metastasis of Colorectal cancer. Surgery is an effective treatment for colorectal cancer with liver metastasis, however, only 10%-20% of patients with liver metastasis are feasible for radical surgical resection.

In the early 1990s, radiofrequency ablation (RFA) was first applied in the treatment of liver metastases. In the late 1990s and early 2000s, microwave ablation (MWA), irreversible electroporation (IRE) and other technologies emerged. Today, with the continuous improvement of ablation techniques, many single-center retrospective studies have demonstrated that thermal ablation for liver metastases is comparable to surgery. Currently, institutions have conducted multi-center randomized controlled trials to compare the outcomes of the two treatment approaches. The expert consensus of tumor ablation therapy has confirmed that the ablation technique has the advantages of minimally invasive, well tolerated and low complications, and has been widely used in the treatment of solid tumors. In the treatment of liver metastases, it also has the advantage of not being limited by residual liver volume.

Postoperative tumor recurrence occurred in about 2/3 of the patients with liver stump, mainly due to the residual microscopic cancer foci. Chemotherapy can kill the microscopic cancer foci of the liver. EORTC (40983) confirmed that: compared with surgery alone, perioperative chemotherapy for resectable liver metastases (<4) could benefit patients with PFS and reduce the incidence of tumor progression-related events. EORTC (40004) proved that in the treatment of non-resectable liver metastases (1 ~ 10, with a maximum diameter <4cm), ablation combined with postoperative chemotherapy was superior to chemotherapy alone. E. Tanis et al compared two randomized controlled trials of EORTC for colorectal cancer liver metastasis, namely 40983 (EPOC) and 40004 (CLOCC), and confirmed the treatment of liver metastasis (<3cm) after integration. There was no significant difference in local recurrence rate between the RFA+ postoperative chemotherapy group and the surgery + perioperative chemotherapy group. At the beginning, neoadjuvant chemotherapy was designed to provide surgical resection opportunities for patients who could not be resected with metastatic tumor. Later, it was gradually applied to resectable liver metastasis. Studies on surgical combination with chemotherapy proved that preoperative chemotherapy was no less effective than postoperative chemotherapy for resectable liver metastasis. However, for isolated small metastatic tumors (<3cm), complete tumor response after neoadjuvant chemotherapy should be avoided, leading to the dilemma of inoperable. Studies have reported that ablation combined with preoperative chemotherapy can cause hepatic steatosis and tumor shrinkage, which makes tumor visualization difficult to a certain extent. If the tumor disappeared on imaging, the pathological specimen confirmed that there were still residues, and the tumor could "reappear" during follow-up. Therefore, the timing of ablation-related chemotherapeutic administration still needs to be explained, and there is still a lack of high-quality evidence-based medical evidence at home and abroad.

The purpose of this study was to compare the clinical efficacy of thermal ablation or combined with perioperative chemotherapy and postoperative chemotherapy in the treatment of colon cancer with liver metastasis.

ELIGIBILITY:
Inclusion Criteria:

* 1) Aged between 18 and 80, WHO physical status score < level 2
* 2) Histologically confirmed colorectal cancer, liver metastasis (≤4), maximum diameter ≤4cm;
* 3) Patients without extrahepatic metastasis;
* 4) If the primary tumor has been resected or has metastasized at the same time, the multidisciplinary panel determines that the primary tumor can be resected and resected within one month after ablation;
* 5) No other chemotherapy experience except anti-tumor treatment for the primary cancer;
* 6) The main organs function normally, that is, they meet the following standards:

  1. Blood routine examination: HB≥90 g/L; The ANC acuity 1.5 x 109 / L; PLT 60 x 109 / L or higher;
  2. Biochemical examination: ALB ≥29g/L; ALT and AST < 3 uln; 1.5 ULN TBIL or less; Creatinine 1.5 or less ULN.

Exclusion Criteria:

* 1) A history of other malignant tumors in the past 5 years;
* 2) Cardiovascular diseases with significant clinical symptoms (uncontrolled congestive heart failure, angina pectoris, hypertension, arrhythmia);
* 3) Persons with coagulation disorders;
* 4) Combined with active infection;
* 5) Those with any contraindications related to chemotherapy;
* 6) Pregnant or lactating women;
* 7) A history of substance abuse and mental illness;
* 8) The investigator believes that there are any other factors that are not suitable for inclusion or affect the subject's participation in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 668 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
DFS | 60 months
  From the beginning of randomization to the time of disease recurrence or death due to disease progression

SECONDARY OUTCOMES:
OS | 60 months
  Time from randomization to death from any cause.
ORR | 60 months
  Proportion of patients whose tumors shrink to a certain extent and remain constant for a certain period of time, including cases of complete response (CR) and partial response (PR).
LTP | 60 months
  From the beginning of randomization to the time of disease progression or death.
CSS | 60 months
  After treatment, death caused by tumor was considered as the end point, and the proportion of patients still alive after several years of follow-up accounted for the total number of follow-up patients.
Tumor reactivity assessment | 60 months
  Tumor reactivity assessment by mRECIST

CONTACTS AND LOCATIONS:
Overall Officials: Ping Liang, Doctor, Principal Investigator — Chinese PLA General Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li J, Pang C, Liu G, Xie X, Zhang DZ, Li K, Li Z, He G, Xu E, Zhong H, Yang H, Lu M, Lou K, Xie X, Lan S, Li Q, Dai G, Yu J, Liang P. Thermal ablation with and without adjuvant systemic therapy: a nationwide multicenter observational cohort study of solitary colorectal liver metastases. Int J Surg. 2024 Jul 1;110(7):4240-4248. doi: 10.1097/JS9.0000000000001397. PMID 38597399